CLINICAL TRIAL: NCT01931566
Title: A Double Blind, Randomized, Placebo Controlled, Parallel Group Study to Simultaneously Qualify a Biomarker Algorithm for Prognosis of Risk of Developing Mild Cognitive Impairment Due to Alzheimer's Disease (MCI Due to AD) and to Test the Safety and Efficacy of Pioglitazone (AD-4833 SR 0.8 mg QD) to Delay the Onset of MCI Due to AD in Cognitively Normal Subjects
Brief Title: Biomarker Qualification for Risk of Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease (AD) and Safety and Efficacy Evaluation of Pioglitazone in Delaying Its Onset
Acronym: TOMMORROW
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy of the drug; no safety concern
Sponsor: Takeda (Industry)
Collaborators: Zinfandel Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD-4833/TOMM40_301; 2012-003111-58 (EudraCT Number); U1111-1139-0355 (Registry Identifier: WHO UTN)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Mild Cognitive Impairment Due to Alzheimer's Disease
Keywords: Drug therapy
MeSH Terms: interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Risk Placebo (Placebo Comparator): Pioglitazone placebo-matching tablets, orally, once daily to participants assigned to low risk group for developing MCI-AD for up to 5 years.
  Interventions: Drug: Pioglitazone placebo
- High Risk Placebo (Placebo Comparator): Pioglitazone placebo-matching tablets, orally, once daily to participants assigned to high risk group for developing MCI-AD for up to 5 years.
  Interventions: Drug: Pioglitazone placebo
- High Risk Pioglitazone (Experimental): Pioglitazone 0.8 mg, sustained release (SR) tablets, orally, once daily to participants assigned to high risk group for developing MCI-AD for up to 5 years.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone SR tablets
  Arms: High Risk Pioglitazone
Drug: Pioglitazone placebo — Pioglitazone placebo-matching tablets
  Arms: High Risk Placebo; Low Risk Placebo

SUMMARY:
The purpose of this study is to qualify the biomarker risk algorithm for prognosis of the risk of developing Mild Cognitive Impairment due to Alzheimer's Disease (MCI-AD), and also to evaluate the efficacy of pioglitazone compared with placebo to delay the onset of MCI-AD in cognitively-normal participants who are at high-risk for developing MCI within 5 years.

DETAILED DESCRIPTION:
This study has two goals. One of these goals is to see if a new genetic test can determine if participants are at risk of developing Mild Cognitive Impairment due to Alzheimer's Disease (MCI-AD) within the next five years. The other goal is to evaluate the study drug called pioglitazone. Pioglitazone is being tested to delay the onset of MCI-AD. This study will look at the effectiveness of pioglitazone in delaying the onset of MCI-AD in cognitively-normal people who are at high-risk of developing MCI-AD, as identified by the biomarker in the non-Hispanic/Latino Caucasian participants.

This multi-centre trial will be conducted worldwide. The study will enroll approximately 3500 subjects. Participants will be assigned to high or low risk groups for developing MCI- AD within the next five years, based on the results of the biomarker risk algorithm. Participants in the high risk group will be randomly assigned to one of the two treatment groups-which will remain unknown to the participant and study doctor during the study (unless there is an urgent medical need):

* Pioglitazone tablet
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

Participants in the low risk group will be assigned to placebo. The assignment of each participant to the high or low risk group, as well as the participant's treatment assignment, will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need).

All participants will be asked to take one tablet at the same time each day throughout the study.

The overall time to participate in this study is approximately 5 years. Participants will make up to 14 visits to the clinic, and will be contacted by telephone 3 months after each treatment visit for a follow-up assessment, and 2 weeks after the final visit.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is able to physically perform the cognitive tests in the opinion of the investigator and is fluent in the language that tests will be administered.
4. Is cognitively normal at baseline, scoring as indicated for the following tests:

   * Clinical Dementia Rating (CDR)=0.
   * At least one memory test above -1.5 standard deviation (SD) of the demographically corrected normative mean.
5. Must score ≥25 on the Mini-Mental State Examination (MMSE) at the screening visit after the education and age adjustment.
6. Is male or postmenopausal female between the ages of 65 and 83 years, inclusive, at time of the Screening visit.
7. Has the ability and intention to participate in regular study visits, in the opinion of the Investigator.
8. Has a project partner who can separately complete an Acknowledgement Form on his/her own behalf and take part in the study (with the intent to do so as long as the participant is enrolled) to provide information on the cognitive, functional, and behavioral status of the participant and to assist with monitoring of study medication, if needed.

Exclusion Criteria:

1. Has a current diagnosis or history of any type of cognitive impairment or dementia or has a current diagnosis or history of neurological/psychiatric disorder or any other diagnosis that significantly affects cognitive performance (eg, mental retardation, organic mental disorder).
2. Has a current diagnosis of significant psychiatric illness, per Diagnostic & Statistical Manual of Mental Disorders, 4th Edition - Text Revision (DSM-IV-TR) (or DSM-V when published) (including but not limited to major depressive disorder, anxiety disorders) and is in an acute phase/episode, or the participant has a current diagnosis or history of schizophrenia or bipolar disorder.
3. Has a glycosylated hemoglobin (HbA1c) >8.0% at the time of baseline or requires treatment with insulin, triple oral antidiabetic therapy or a peroxisome proliferator-activated receptor-gamma (PPAR-γ) agonist. The participant should be on a stable antidiabetic regimen for at least 3 months prior to enrollment.
4. Has a clinically significant unstable illness, for example, hepatic impairment or renal insufficiency, or cardiovascular, pulmonary, gastrointestinal (including s/p gastric bypass), endocrine, neurological, rheumatologic, immunologic, infectious, skin and subcutaneous tissue disorders, or metabolic disturbance. History of HIV infection is considered exclusionary for this study.
5. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse/dependence within 2 years prior to the Screening Visit.
6. Is an immediate family member, testing center employee, or is in a dependent relationship with a testing center employee who is involved in conduct of this study (eg, spouse, parent, child, and sibling) or may consent under duress.
7. Has a history of hypersensitivity or allergies to pioglitazone or related compounds.
8. Is required to take excluded medications as specified in the Excluded Medications Section.
9. Had any of the following values at the Baseline Visit (Visit 2):

   1. A serum total bilirubin value >1.5× upper limit of normal (ULN).
   2. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2xULN.
   3. Unexplained microscopic/macroscopic hematuria on one repeat examinations within 2 weeks of the initial assessment.
10. Is positive for either Hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV) antibodies at the Baseline Visit (Visit 2).
11. Has a condition or takes medication that, in the opinion of the Investigator, could interfere with the assessments of safety, tolerability, or efficacy, or prevent the participant from adequately participating in the study or continue for the anticipated duration of the study.
12. Has received any investigational compound within 30 days prior to screening or 5 half-lives prior to Screening or is currently participating in another study which entails the administration of an investigational or marketed drug, supplement or intervention including, but not limited to diet, exercise, lifestyle or invasive procedure.
13. Has a history of any cancer that has been in remission for less than 2 years from the Screening Visit. Participants with basal cell or stage I squamous cell carcinoma of the skin will be eligible. Participants with history of bladder cancer are not eligible irrespective of the remission status.
14. Has a history or current diagnosis of macular edema or macular degeneration.
15. If female, has a history of postmenopausal fractures with no or minimal trauma (eg, wrist, hip, lumbar or thoracic vertebral fracture).
16. Has a history or current diagnosis of congestive heart failure (CHF), New York Heart Association Class III-IV.
17. Has been exposed to the cognitive tests performed in this study within 6 months prior to the Screening Visit, with the exception of the MMSE.
18. Participant's Translocase of the Outer Mitochondrial Membrane 40 homolog (TOMM40) rs10524523 or apolipoprotein E (APOE) genotypes or APOE phenotype are known by the participant or the study staff participating in this study.

Ages: 65 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 3494 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (55):
- United States (34):
  - Phoenix, Arizona
  - Sun City, Arizona
  - Long Beach, California
  - San Diego, California
  - San Francisco, California
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Lady Lake, Florida
  - Lake Worth, Florida
  - Merritt Island, Florida
  - Orlando, Florida
  - Port Orange, Florida
  - St. Petersburg, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Elk Grove, Illinois
  - Elk Grove Village, Illinois
  - Iowa City, Iowa
  - Farmington Hills, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Marlton, New Jersey
  - New York, New York
  - Concord, North Carolina
  - Durham, North Carolina
  - Akron, Ohio
  - Portland, Oregon
  - Charleston, South Carolina
  - Cordova, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Middleton, Wisconsin
- Australia (4):
  - North Ryde, New South Wales
  - Southport, Queensland
  - West Heidelberg, Victoria
  - Nedlands, Western Australia
- Germany (4):
  - Stuttgart, Baden-Wurttemberg
  - Siegen, North Rhine-Westphalia
  - Halle, Saxony-Anhalt
  - Berlin
- Basel, Switzerland
- United Kingdom (12):
  - Exeter, Devon
  - Plymouth, Devon
  - Hammersmith, Greater London
  - London, Greater London
  - Manchester, Greater Manchester
  - Salford, Greater Manchester
  - Blackpool, Lancashire
  - Isleworth, Middlesex
  - Glasgow, Strathclyde
  - Dundee, Tayside Region
  - Perth, Tayside Region
  - Bristol

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Zou H, Luo S, Liu H, Lutz MW, Bennett DA, Plassman BL, Welsh-Bohmer KA. Genotypic Effects of the TOMM40'523 Variant and APOE on Longitudinal Cognitive Change over 4 Years: The TOMMORROW Study. J Prev Alzheimers Dis. 2023;10(4):886-894. doi: 10.14283/jpad.2023.115. PMID 37874111
- [Derived] Burns DK, Alexander RC, Welsh-Bohmer KA, Culp M, Chiang C, O'Neil J, Evans RM, Harrigan P, Plassman BL, Burke JR, Wu J, Lutz MW, Haneline S, Schwarz AJ, Schneider LS, Yaffe K, Saunders AM, Ratti E; TOMMORROW study investigators. Safety and efficacy of pioglitazone for the delay of cognitive impairment in people at risk of Alzheimer's disease (TOMMORROW): a prognostic biomarker study and a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2021 Jul;20(7):537-547. doi: 10.1016/S1474-4422(21)00043-0. PMID 34146512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 57 investigative sites in United States, United Kingdom, Germany, Australia, and Switzerland from 01 Aug 2013 to 06 Sep 2018.
Pre-assignment Details: Participants at least 65 years old with normal cognitive function were enrolled to receive either pioglitazone (0.8 mg sustained release tablet) or placebo.
Period: Overall Study
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone
Started | 433 | 1516 | 1545
Treated | 427 | 1507 | 1531
Completed (Completed here refers to those participants who completed study drug.) | 4 | 40 | 39
Not Completed | 429 | 1476 | 1506
Not completed — Randomized But Not Treated | 6 | 9 | 14
Not completed — Adverse Event | 37 | 167 | 132
Not completed — Major Protocol Deviation | 5 | 14 | 21
Not completed — Lost to Follow-up | 3 | 26 | 23
Not completed — Voluntary Withdrawal | 78 | 245 | 225
Not completed — Study Termination | 289 | 968 | 1037
Not completed — Reason Not Specified | 11 | 47 | 53
Not completed — Missing | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone | Total
Number analyzed (Participants) | 433 | 1516 | 1545 | 3494
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (4.02) | 74.6 (5.27) | 74.4 (5.25) | 74.0 (5.31)
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 360 | 632 | 658 | 1650
  >=75 years | 73 | 884 | 887 | 1844
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 850 | 812 | 1921
  Male | 174 | 666 | 733 | 1573
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 19 | 12 | 39
  Not Hispanic or Latino | 425 | 1497 | 1533 | 3455
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 4 | 4
  Asian | 1 | 10 | 14 | 25
  Black or African American | 10 | 38 | 39 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  White | 421 | 1463 | 1484 | 3368
  Multiracial | 1 | 4 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic/Latino Caucasian | 413 | 1444 | 1472 | 3329
  Hispanic/Latino and/or non-Caucasian | 20 | 72 | 73 | 165
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 270 | 962 | 985 | 2217
  United Kingdom | 102 | 311 | 315 | 728
  Australia | 56 | 215 | 218 | 489
  Switzerland | 3 | 18 | 18 | 39
  Germany | 2 | 10 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Time to Diagnosis of Mild Cognitive Impairment Due to Alzheimer's Disease (MCI-AD) for Placebo-treated, High-risk, Non-Hispanic/Latino Caucasian Participants Versus Placebo-treated, Low-risk, Non-Hispanic/Latino Caucasian Participants
Description: The event definition for MCI-AD was the time in days from the randomization date to the date of the first of two consecutive scheduled visits at which a participant was assessed with a diagnosis of MCI due to AD confirmed by adjudication committee. Here, the time to event was reported as the restricted mean survival time. The restricted mean survival time was defined as the area under the curve of the survival function up to the largest event time.
Time Frame: Baseline to the end of study (approximately up to 5 years)
Population: Full Analysis Set (FAS) included all participants who were randomized, received at least 1 dose of study drug, and at least 1 valid postbaseline value for assessment of primary efficacy. A participant who does not have an event of MCI due to AD was censored at the date of the last visit at which MCI due to AD could have been assessed.
Measure: Mean (Full Range); unit: days
Arm/Group | Low Risk Placebo | High Risk Placebo
Number analyzed (Participants) | 402 | 1406
days | 905.44 [189.00 to 909.00] | 1238.67 [168.00 to 1268.00]
Statistical Analysis 1: Comparison: Low Risk Placebo vs High Risk Placebo; Test type: Other; p = 0.023, Regression, Cox

2. Primary Outcome: Time to Diagnosis of MCI Due to AD for Pioglitazone-treated, High-risk, Non-Hispanic/Latino Caucasian Participants Versus Placebo-treated, High-risk, Non-Hispanic/Latino, Caucasian Participants
Description: as for outcome 1
Time Frame: Baseline to the end of study (approximately up to 5 years)
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and at least 1 valid postbaseline value for assessment of primary efficacy. A participant who does not have an event of MCI due to AD was censored at the date of the last visit at which MCI due to AD could have been assessed.
Measure: Mean (Full Range); unit: days
Arm/Group | High Risk Placebo | High Risk Pioglitazone
Number analyzed (Participants) | 1406 | 1430
days | 1238.67 [168.00 to 1268.00] | 1261.24 [168.00 to 1285.00]
Statistical Analysis 1: Comparison: High Risk Placebo vs High Risk Pioglitazone; Test type: Superiority; p = 0.307, Regression, Cox

3. Secondary Outcome: Change From Baseline for Cognitive Decline on Composite Score on the Cognitive Test Battery for Pioglitazone-treated Participants Versus Placebo-treated Participants in the High-risk Stratum
Description: Composite scores derived from the test battery. Domains of Episodic Memory [California Verbal Learning Test-2nd Edition (CVLT-II), Brief Visuospatial Memory Test-Revised (BVMT-R)]; Executive Function [Trail Making Test (TMT) (Part B), Wechsler Adult Intelligence Scale (WAIS)-III Digit Span Test-backwards span]; Language [Multilingual Naming Test (MiNT), Semantic Fluency (animals), Lexical/phonemic fluency (F, A, and S in English; D, S, and F in German)]; and Attention [WAIS-III Digit Span Test-forward span, TMT (Part A)] used for composite score. 12 measures were derived from 8 neuropsychological tests. CVLT-II test involved 2 primary measures (short, long delay recall); BVMT-R had 2 measures (copy and recall); Digit Span and Trail both had 2 measures (forward and backward span and Parts A and B). There was 1 total score for each test: CDT, MINT, semantic and lexical fluency. Total score ranged from -1.222 to 1.707 at baseline, a higher composite score indicated better cognition.
Time Frame: Baseline and Month 48
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and at least 1 valid postbaseline value for assessment of primary efficacy. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk Placebo | High Risk Pioglitazone
Number analyzed (Participants) | 1406 | 1430
score on a scale | 0.1841 (0.27508) | 0.1687 (0.40621)

4. Secondary Outcome: Change From Baseline in Instrumental Activities of Daily Living (Alzheimer's Disease Cooperative Study Activities of Daily Living - Prevention Instrument [ADCS ADL-PI]) Between Pioglitazone-treated and Placebo-treated Groups of the High-risk Stratum
Description: The ADCS ADL-PI is a functional measure that was specifically designed for standardized administration over long duration clinical studies to prevent AD. The ADCS ADL-PI is a 20-item instrument that included 15 ADL questions, which were scored as 1 (with a lot of difficulty), 2 (with some difficulty), or 3 (as well as usually, with no difficulty), plus 5 vision, hearing, and mobility questions, which were scored from 0 (no) to 1 (yes). ADL Total ranged from 0 to 45, and lower scores indicated greater disability.
Time Frame: Baseline and Month 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk Placebo | High Risk Pioglitazone
Number analyzed (Participants) | 1406 | 1430
score on a scale | 0.1 (4.93) | 0.3 (5.32)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study drug (up to 935 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone
All-Cause Mortality (participants affected / at risk) | 2/427 | 21/1507 | 7/1531
Serious Adverse Events (participants affected / at risk) | 81/427 | 404/1507 | 358/1531
Other Adverse Events (participants affected / at risk) | 235/427 | 828/1507 | 822/1531
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk Placebo (N=427) | High Risk Placebo (N=1507) | High Risk Pioglitazone (N=1531)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 15 | 16
Angina pectoris (Cardiac disorders) | 3 | 10 | 6
Coronary artery disease (Cardiac disorders) | 2 | 7 | 7
Myocardial infarction (Cardiac disorders) | 0 | 13 | 3 — Four treatment-emergent deaths occurred during treatment with placebo (in high-risk group) and were not related.
Cardiac failure congestive (Cardiac disorders) | 1 | 8 | 6 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was related. One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Acute myocardial infarction (Cardiac disorders) | 1 | 5 | 3 — One treatment-emergent death occurred during treatment with pioglitazone (in high-risk group) and was not related.
Sinus node dysfunction (Cardiac disorders) | 0 | 2 | 5
Bradycardia (Cardiac disorders) | 0 | 4 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 5
Cardiac arrest (Cardiac disorders) | 0 | 3 | 2 — Two treatment-emergent deaths occurred during treatment with placebo (in high-risk group) and were not related.
Ventricular tachycardia (Cardiac disorders) | 1 | 3 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 2 | 1
Angina unstable (Cardiac disorders) | 0 | 3 | 0
Arrhythmia (Cardiac disorders) | 0 | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 1 — One treatment-emergent death occurred during treatment with pioglitazone (in high-risk group) and was not related.
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 1
Extrasystoles (Cardiac disorders) | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 1
Atrial septal defect acquired (Cardiac disorders) | 0 | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Congenital cerebrovascular anomaly (Congenital, familial and genetic disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 3
Vertigo positional (Ear and labyrinth disorders) | 1 | 3 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 2 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 5
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 4
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gallstone ileus (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 5 | 8
Asthenia (General disorders) | 0 | 0 | 2
Chest pain (General disorders) | 0 | 2 | 0
Hernia (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Fatigue (General disorders) | 0 | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Unevaluable event (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 3 | 6
Cholecystitis acute (Hepatobiliary disorders) | 0 | 3 | 3
Cholelithiasis (Hepatobiliary disorders) | 2 | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Primary biliary cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 12 | 15 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Diverticulitis (Infections and infestations) | 3 | 7 | 4
Cellulitis (Infections and infestations) | 1 | 3 | 8
Sepsis (Infections and infestations) | 1 | 5 | 6
Urosepsis (Infections and infestations) | 2 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 5 | 3
Appendicitis (Infections and infestations) | 2 | 1 | 4
Gastroenteritis (Infections and infestations) | 0 | 3 | 4
Lower respiratory tract infection (Infections and infestations) | 1 | 2 | 3
Influenza (Infections and infestations) | 0 | 4 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 2 | 1
Wound infection (Infections and infestations) | 1 | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 7 | 3
Hip fracture (Injury, poisoning and procedural complications) | 2 | 7 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 4 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 4 | 1 — Two treatment-emergent deaths occurred during treatment with placebo (in high-risk group) and were not related.
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 3 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 3 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 3
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Periprosthetic osteolysis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Flatback syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 — One treatment-emergent death occurred in participant who also suffered from cerebrovascular accident during treatment with placebo (in high-risk group) and was not related.
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Blood parathyroid hormone increased (Investigations) | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 22 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 13 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8 | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1 — One treatment-emergent death occurred during treatment with placebo (in low-risk group) and was not related. Two treatment-emergent deaths occurred during treatment with placebo (in high-risk group) and were not related.
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 — One treatment-emergent death occurred during treatment with pioglitazone (in high-risk group) and was not related.
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with pioglitazone (in high-risk group) and was not related.
Choroid plexus papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intracranial meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mucinous breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was related.
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with pioglitazone (in high-risk group) and was not related.
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 13 | 14
Transient ischaemic attack (Nervous system disorders) | 0 | 11 | 10
Cerebrovascular accident (Nervous system disorders) | 1 | 10 | 6 — One treatment-emergent death occurred in participant who also suffered from subdural haemorrhage during treatment with placebo (in high-risk group) and was not related.
Presyncope (Nervous system disorders) | 1 | 4 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 3 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 3
Cerebral haemorrhage (Nervous system disorders) | 0 | 3 | 0 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Seizure (Nervous system disorders) | 1 | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 2 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Facial neuralgia (Nervous system disorders) | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Temporal lobe epilepsy (Nervous system disorders) | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 5 | 7
Urinary retention (Renal and urinary disorders) | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urinoma (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 4 | 2
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 11
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 — One treatment-emergent death occurred during treatment with placebo (in high-risk group) and was not related.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 — One treatment-emergent death occurred during treatment with pioglitazone (in high-risk group) and was not related.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 — One treatment-emergent death occurred during treatment with pioglitazone (in high-risk group) and was not related.
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 3 | 2
Hypotension (Vascular disorders) | 1 | 4 | 1 — One treatment-emergent death occurred during treatment with placebo (in low-risk group) and was not related.
Aortic stenosis (Vascular disorders) | 0 | 3 | 2
Aortic aneurysm (Vascular disorders) | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 1 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 1
Varicose vein (Vascular disorders) | 0 | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Superior mesenteric artery syndrome (Vascular disorders) | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk Placebo (N=427) | High Risk Placebo (N=1507) | High Risk Pioglitazone (N=1531)
Cataract (Eye disorders) | 27 | 119 | 106
Constipation (Gastrointestinal disorders) | 24 | 70 | 72
Upper respiratory tract infection (Infections and infestations) | 62 | 190 | 183
Urinary tract infection (Infections and infestations) | 47 | 178 | 191
Nasopharyngitis (Infections and infestations) | 22 | 72 | 90
Sinusitis (Infections and infestations) | 22 | 67 | 52
Fall (Injury, poisoning and procedural complications) | 18 | 143 | 135
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 125 | 125
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 82 | 101
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 81 | 86
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 | 59 | 71
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 79 | 76
Hypertension (Vascular disorders) | 26 | 97 | 93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT01931566/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT01931566/SAP_001.pdf